CLINICAL TRIAL: NCT01198639
Title: One-year Mortality According to the Method of Total Intravenous Anesthesia. A Prospective, Randomized and Multicenter Study
Brief Title: One-year Mortality After Surgery and Low Bispectral Index
Acronym: ELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/30
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- manual administration of iv anesthetics (Active Comparator)
  Interventions: Device: manual administration of iv anesthetics (propofol and remifentanil) using the Toolbox platform
- closed-loop administration of iv anesthetics (Experimental)
  Interventions: Device: closed-loop administration of iv anesthetics (propofol and remifentanil) using the Toolbox platform

INTERVENTIONS:
Device: manual administration of iv anesthetics (propofol and remifentanil) using the Toolbox platform — the anesthesiologists are instructed to maintain the BIS values between 40 and 60 throughout anesthesia using target controlled infusion method
  Arms: manual administration of iv anesthetics
Device: closed-loop administration of iv anesthetics (propofol and remifentanil) using the Toolbox platform — an algorithm is used to maintain automatically the BIS values between 40 and 60
  Arms: closed-loop administration of iv anesthetics

SUMMARY:
A correlation between deep anesthesia (defined as time with Bispectral Index (BIS) lower than 45) and death within 1 yr after surgery has previously been reported. In order to confirm or refute these findings, the investigators have designed a study which compares two methods of administration for total intravenous anesthesia (propofol and remifentanil):

* manual administration: the anesthesiologists are instructed to maintain the BIS value between 40 and 60.
* closed loop administration: an algorithm is used to maintain the BIS value between 40 and 60.

Based on previous studies, the amount of time that BIS is maintained above 40 is greater when anesthetics agents are administered using closed loop compared with manual administration.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology patient classification status I, II and III
* patients aged between 50 and 85 years old
* born in France
* surgical procedures lasting more than one hour

Exclusion Criteria:

* American Society of Anesthesiology patient classification status IV
* patients born out of France
* pace-maker
* surgical procedure on the skull or avoiding an adequate positioning of the bispectral index electrode dementia, history of central nervous system disease (tumor, vascular event, Parkinson disease, ...)
* psychiatric illness (severe depression or psychosis), patients receiving a psychotropic treatment
* anesthesia performed during the year before inclusion in this study except for diagnostic procedures
* allergy to propofol, soja, peanuts, or to sufentanil, remifentanil, or morphine, to a myorelaxant or to an excipient,
* hypersensibility to sufentanil, to remifentanil, or to other derivate of fentanyl

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2044 (Actual)
Dates: Start 2010-09-13 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Mortality rate during the first year following anesthesia | one year after anesthesia

SECONDARY OUTCOMES:
conduct of anesthesia (duration of anesthesia with bispectral index < 45, bispectral index < 40, bispectral index > 60, bispectral index > 65, and burst suppression ratio) | end of anesthesia
intraoperative awareness | one month postoperatively
patients' satisfaction in the postanesthesia care unit (nausea, vomiting, shivering) | end of the stay in the postanesthesia care unit
postoperative complication during the hospital stay (ancillary study) | one month after anesthesia
major medical events during the first year following anesthesia | one year after anesthesia
relation between patients' characteristics and mortality rate during the first year following anesthesia | one year after anesthesia
intraoperative parameters, notably hemodynamic parameters, and their relation between them and mortality rate during the first year following anesthesia | one year after anesthesia
in-hospital and one month mortality | one year after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (22):
- France (22):
  - CHU Victor Dupuy, Argenteuil
  - CHU Besançon, Besançon
  - Hôpitaux Universitaires Paris-Seine St Denis CHU Avicenne, Bobigny
  - Clinique Saint Augustin, Bordeaux
  - Clinique Saint Vincent de Paul, Bourgoin
  - Hôpital Femme-Mère-Enfant, Bron
  - CH de Chartres Louis Pasteur, Chartres
  - H.I.A Percy, Clamart
  - Centre Jean Perrin, Clermont-Ferrand
  - Clinique des Deux Caps, Coquelles
  - Clinique Fontaine-lès-Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Institut Hospitalier Franco Britannique, Levallois-Perret
  - Institut Paoli-Calmettes, Marseille
  - HIA du Val de Grace, Paris
  - HEGP, Paris
  - CHI Poissy/St Germain-en-Laye, Poissy
  - CHU de Rouen, Rouen
  - Hia Begin, Saint-Mandé
  - Hôpital Foch, Suresnes
  - CHU Rangueil, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Background] Cantraine FR, Coussaert EJ. The first object oriented monitor for intravenous anesthesia. J Clin Monit Comput. 2000 Jan;16(1):3-10. doi: 10.1023/a:1009904805940. PMID 12578088
- [Result] Lindholm ML, Traff S, Granath F, Greenwald SD, Ekbom A, Lennmarken C, Sandin RH. Mortality within 2 years after surgery in relation to low intraoperative bispectral index values and preexisting malignant disease. Anesth Analg. 2009 Feb;108(2):508-12. doi: 10.1213/ane.0b013e31818f603c. PMID 19151279
- [Result] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Derived] Mahr N, Bouhake Y, Chopard G, Liu N, Boichut N, Chazot T, Claveau M, Vettoretti L, Tio G, Pili-Floury S, Samain E, Besch G. Postoperative Neurocognitive Disorders After Closed-Loop Versus Manual Target Controlled-Infusion of Propofol and Remifentanil in Patients Undergoing Elective Major Noncardiac Surgery: The Randomized Controlled Postoperative Cognitive Dysfunction-Electroencephalographic-Guided Anesthetic Administration Trial. Anesth Analg. 2021 Oct 1;133(4):837-847. doi: 10.1213/ANE.0000000000005278. PMID 33181558